CLINICAL TRIAL: NCT03929133
Title: Development of an Screening System in Children With Congenital Heart Disease Based on Cloud Computing and Big Data
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-16-040
Record Dates: First submitted 2016-11-22; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2018-12

CONDITIONS: Heart Diseases
Keywords: fetal heart sounds; big data; cloud computing; congenital heart disease; data base; Acoustic structure design
MeSH Terms: conditions — Heart Diseases; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: automatic screening machine on congenital heart disease

SUMMARY:
This study intends to establish an automatic system for screening on children with congenital heart disease, the system include the auscultation of cardiac murmur and the test of oxygen saturation, the data was analyzed based on the cloud computing.

DETAILED DESCRIPTION:
This study intends to establish a system for screening of children with congenital heart disease,with the combination of cardiac auscultation , the test of oxygen saturation, the use of cloud computing and data base. The investigators decide to do this project from three main points.1:How to establish a data-base system? 2:How to get heart sound signal? 3.How to analyze so many signals?

ELIGIBILITY:
Inclusion Criteria:

* Neonatal ward patients
* Patients with echocardiography reports

Exclusion Criteria:

* Severe pneumonia

Max Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study include between between newborn to 10 years old.Heart sound signal need to be collected to analyze children's heart health status and creat a special model of each kind of CHD.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value | 2days
  The ratio of truly congenital heart disease cases divide by the total positive cases detected by the screening test.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Pengjun, MD, Study Director — Pediatric cardiovascular department, Shanghai xinhua hospital
Locations (1):
- Zhao Pengjun, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The investigator do not plan to share the data until the project is totally completed

REFERENCES:
- [Background] van der Linde D, Konings EE, Slager MA, Witsenburg M, Helbing WA, Takkenberg JJ, Roos-Hesselink JW. Birth prevalence of congenital heart disease worldwide: a systematic review and meta-analysis. J Am Coll Cardiol. 2011 Nov 15;58(21):2241-7. doi: 10.1016/j.jacc.2011.08.025. PMID 22078432
- [Background] Ho TC, Ouyang H, Lu Y, Young AH, Chintala K, Detrano RC. Postprocedural outcomes of rural children undergoing correction of congenital heart lesions in Yunnan Province, China. Pediatr Cardiol. 2011 Aug;32(6):811-4. doi: 10.1007/s00246-011-9991-y. Epub 2011 Apr 11. PMID 21479905
- [Background] Zhao QM, Ma XJ, Ge XL, Liu F, Yan WL, Wu L, Ye M, Liang XC, Zhang J, Gao Y, Jia B, Huang GY; Neonatal Congenital Heart Disease screening group. Pulse oximetry with clinical assessment to screen for congenital heart disease in neonates in China: a prospective study. Lancet. 2014 Aug 30;384(9945):747-54. doi: 10.1016/S0140-6736(14)60198-7. Epub 2014 Apr 22. PMID 24768155
- [Background] G. Douglas et al., Macleod's Clinical Examination. New York, NY, USA: Elsevier Health Sciences, 2009
- [Background] A. G. Tilkian and M. B. Conover, Understanding Heart Sounds and Murmurs: With an Introduction to Lung Sounds.NewYork,NY, USA: ElsevierHealth Sciences, 2001.
- [Background] KUN-HIS TSAI. METHOD, SYSTEM AND DEVICE FOR AUSCULTATION：US，US2016/0143612 A1[P]. 2016
- [Background] Barry Poplaw. PORTABLE SMART STETHOSCOPE FORMED OF SMART MOBILE DEVICE AND CASING ASSEMBLY：US，US 2015/0327812 A1[P]. 2015
- [Background] Winther S, Schmidt SE, Holm NR, Toft E, Struijk JJ, Botker HE, Bottcher M. Diagnosing coronary artery disease by sound analysis from coronary stenosis induced turbulent blood flow: diagnostic performance in patients with stable angina pectoris. Int J Cardiovasc Imaging. 2016 Feb;32(2):235-245. doi: 10.1007/s10554-015-0753-4. Epub 2015 Sep 3. PMID 26335368
- [Background] Visagie C, Scheffer C, Lubbe WW, Doubell AF. Autonomous detection of heart sound abnormalities using an auscultation jacket. Australas Phys Eng Sci Med. 2009 Dec;32(4):240-50. doi: 10.1007/BF03179245. PMID 20169844
- [Background] Huang GY. Screening markers of congenital heart disease and their clinical values. Chinese Journal of Practical Pediatrics , 2013(7):503-504
- [Background] Zhang HX,Cheng XF.Heart sound analysis virtual instrument based on LabVIEW platform. Computer Technology and Development,2010,11:217-220